CLINICAL TRIAL: NCT05099055
Title: Dexmedetomidine Comme Adjuvant à la rachianesthésie Lors de césariennes électives : Une étude Pilote
Brief Title: Dexmedetomine as Adjuvant for Spinal Anesthesia in Elective Cesarian Sections : a Pilot Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Christina Lamontagne, Anesthesioligist, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-3543
Record Dates: First submitted 2021-10-17; First posted 2021-10-29 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Analgesia; Analgesics, Opioid; Anesthesia, Obstetrical; Anesthesia, Spinal; Analgesics, Non-Narcotic; Dexmedetomidine; Analgesia, Obstetrical
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine; Analgesics, Opioid

STUDY DESIGN:
Intervention Model Description: Pilot study for a phase 3 study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (Experimental): Monitoring will be installed upon arrival.Metoclopramide 10 mg IV and Dexamethasone 4 mg will be given for nausea-prophylaxis. Patients may be given ondansetron 4 mg as rescue. Cefazoline 2G or clindamycin 900 mg will be given.A sterile spinal technique will be performed with a 25G Whitacre. Bupivacaine 12 mg (1.6 ml) will be drawn and given, along with dexmedetomidine 3 mcg (0.75 mL) previously blindly prepared for a total of 2.35 ml.Adequate blood pressure will be maintained with phenylephrine infusion or ephedrine IV. Glycopyrrolate 0.2 mg may be given for bradycardia.Once an adequate sensory block is obtained, the obstetrics team can perform the surgery.The patient will receive a dose of ketorolac 30 mg IV before leaving the PACU and then Naproxen 500 mg PO every 12 hours.She will receive acetaminophen 975 mg PO every 6 hours and hydromorphone 2-4 mg PO every 3 hours prn. Patients will also have access to a protocol for treatment of nausea and pruritus.
  Interventions: Drug: Dexmedetomidine 0.004 MG/ML [Precedex]
- Control group (Active Comparator): Monitoring will be installed upon arrival.Metoclopramide 10 mg IV and Dexamethasone 4 mg will be given for nausea-prophylaxis. Patients may be given ondansetron 4 mg as rescue. Cefazoline 2G or clindamycin 900 mg will be given.A sterile spinal technique will be performed with a 25G Whitacre. Bupivacaine 12 mg (1.6 ml) will be drawn and given, along with morphine 100 mcg, fentanyl 15 mcg and normal saline 0.25 ml previously blindly prepared for a total of 2.35 ml.Adequate blood pressure will be maintained with phenylephrine infusion or ephedrine IV. Glycopyrrolate 0.2 mg may be given for bradycardia.Once an adequate sensory block is obtained, the obstetrics team can perform the surgery.The patient will receive a dose of ketorolac 30 mg IV before leaving the PACU and then Naproxen 500 mg PO every 12 hours.She will receive acetaminophen 975 mg PO every 6 hours and hydromorphone 2-4 mg PO every 3 hours prn. Patients will also have access to a protocol for treatment of nausea and pruritus.
  Interventions: Drug: Opioids

INTERVENTIONS:
Drug: Dexmedetomidine 0.004 MG/ML [Precedex] — Injection of 3 mcg of dexmedetomidine and 12 mg of bupivacaine in the intrathecal space to provide spinal anesthesia.
  Arms: Test group
Drug: Opioids — Injection of 100 mcg of morphine, 15 mcg of fentanyl and 0.25 ml of normal salin (sterile) with 12 mg of bupivacaine in the intrathecal space to provide spinal anesthesia.
  Arms: Control group

SUMMARY:
The proposed pilot study is a prospective, randomized, controlled, double-blind, single-center pilot study.The aim of this pilot project is to evaluate the feasibility of a phase III study on the use of dexmedetomidine in intrathecal in the context of elective cesarean section.

The target population for the study will be adult pregnant women undergoing elective cesarean section under spinal anesthesia. This study will be carried out at a single site, the CHU Sainte-Justine as part of a research internship as part of the anesthesiology residency program at the University of Montreal.

DETAILED DESCRIPTION:
52 patients will be recruted for this study, and will be randomized in two equal groups.

All the interventions carried out will be standardized. Medical care for patients will be the same as usual care, except for administration of dexmedetomidine or intrathecal narcotics.

In the test group, bupivacaine (12 mg, 1.6 ml) will be injected with 3 mcg of dexemedetomidine.

In the second group, bupivacaine (12 mg, 1.6 ml) will be injected with 100 mcg of morphine and 15 mcg of fentanyl with 0.25 ml of normal saline, which corresponds to the standard treatment.

The patients will receive standard analgesia, described in the protocol, post-operatively and will also have access to anti-nausea and anti-pruritics.

The patient will then be seen the day after surgery to collect her validated self-assessment scales for pain, nausea and vomiting, pruritus, chills and complete her QoR15 questionnaire.

This will be collected to establish preliminary data for a second study of non-inferiority for analgesia and gradation of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patient will receive an elective c-section under spinal anesthesia
* Gestational age > 37 weeks

Exclusion Criteria:

* ASA score ≥ 3
* Allergy or contraindication to receiving opioids (morphine or fentanyl)
* Allergy or contraindication to receiving anti-inflammatory drugs (ketorolac, Naprosyn)
* Allergy or contraindication to receiving acetaminophen
* Height <152 cm or> 183 cm
* Weight <50 or> 110 kg
* Contraindication to spinal anesthesia
* Conversion to general anesthesia
* Combined spinal-epidural anesthesia
* Inability to give informed consent, either secondary to a mental or physical disability or a significant language barrier (Inability to understand English or French)
* Need for transfusion or other major complication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Phase 3 study feasability | 3 months
  The primary outcome will be to evaluate the phase 3 study feasability through recrutement rates and time needed to recrut a total of 52 patients

SECONDARY OUTCOMES:
Opioids consumption | 24 hours post-operatively
  Total morphine equivalent consumed by the patient
Pruritus | 2, 6, 12 and 24 hours after surgery
  Self-assessed validated numerical pruritus scale (NPS). Scale between 0 and 10, 10 being the worst symptoms the patient can imagine.
Nausea | 2, 6, 12 and 24 hours after surgery
  Absence or presence of nausea / vomiting at 2, 6, 12 and 24 hours after surgery
Pain level | 2, 6, 12 and 24 hours after surgery
  Self-assessed validated numerical pain scale (NPS).Scale between 0 and 10, 10 being the worst symptoms the patient can imagine.
Quality of recovery and patient's satisfaction | 24 hours after surgery
  Satisfaction according to the QoR15 questionnaire. Questionnaire containing 15 question to evaluate the quality of recovery in patients after a surgery.
Nausea | 24 hours post-operatively
  Number of anti-nausea medication doses needed

CONTACTS AND LOCATIONS:
Overall Officials: Christina Lamontagne, Study Director — Ste-Justine's Hospital
Locations (1):
- Ste-Justine Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gu J, Karmakar-Hore S, Hogan ME, Azzam HM, Barrett JFR, Brown A, Cook JL, Jain V, Melamed N, Smith GN, Zaltz A, Gurevich Y. Examining Cesarean Section Rates in Canada Using the Modified Robson Classification. J Obstet Gynaecol Can. 2020 Jun;42(6):757-765. doi: 10.1016/j.jogc.2019.09.009. Epub 2019 Dec 26. PMID 31883751
- [Background] Menacker F, Hamilton BE. Recent trends in cesarean delivery in the United States. NCHS Data Brief. 2010 Mar;(35):1-8. PMID 20334736
- [Background] American Society of Anesthesiologists Task Force on Obstetric Anesthesia. Practice guidelines for obstetric anesthesia: an updated report by the American Society of Anesthesiologists Task Force on Obstetric Anesthesia. Anesthesiology. 2007 Apr;106(4):843-63. doi: 10.1097/01.anes.0000264744.63275.10. No abstract available. PMID 17413923
- [Background] Palmer CM, Emerson S, Volgoropolous D, Alves D. Dose-response relationship of intrathecal morphine for postcesarean analgesia. Anesthesiology. 1999 Feb;90(2):437-44. doi: 10.1097/00000542-199902000-00018. PMID 9952150
- [Background] Dahl JB, Jeppesen IS, Jorgensen H, Wetterslev J, Moiniche S. Intraoperative and postoperative analgesic efficacy and adverse effects of intrathecal opioids in patients undergoing cesarean section with spinal anesthesia: a qualitative and quantitative systematic review of randomized controlled trials. Anesthesiology. 1999 Dec;91(6):1919-27. doi: 10.1097/00000542-199912000-00045. No abstract available. PMID 10598635
- [Background] Chaney MA. Side effects of intrathecal and epidural opioids. Can J Anaesth. 1995 Oct;42(10):891-903. doi: 10.1007/BF03011037. PMID 8706199
- [Background] Goldberg RF. The Opioid Crisis: The Surgeon's Role. Adv Surg. 2019 Sep;53:305-325. doi: 10.1016/j.yasu.2019.04.015. Epub 2019 May 17. No abstract available. PMID 31327454
- [Background] Volkow ND, Blanco C. The changing opioid crisis: development, challenges and opportunities. Mol Psychiatry. 2021 Jan;26(1):218-233. doi: 10.1038/s41380-020-0661-4. Epub 2020 Feb 4. PMID 32020048
- [Background] Coussens NP, Sittampalam GS, Jonson SG, Hall MD, Gorby HE, Tamiz AP, McManus OB, Felder CC, Rasmussen K. The Opioid Crisis and the Future of Addiction and Pain Therapeutics. J Pharmacol Exp Ther. 2019 Nov;371(2):396-408. doi: 10.1124/jpet.119.259408. Epub 2019 Sep 3. PMID 31481516
- [Background] Pan PH. Post cesarean delivery pain management: multimodal approach. Int J Obstet Anesth. 2006 Jul;15(3):185-8. doi: 10.1016/j.ijoa.2006.04.004. No abstract available. PMID 16798441
- [Background] Li R, Qi F, Zhang J, Ji Y, Zhang D, Shen Z, Lei W. Antinociceptive effects of dexmedetomidine via spinal substance P and CGRP. Transl Neurosci. 2015 Dec 16;6(1):259-264. doi: 10.1515/tnsci-2015-0028. eCollection 2015. PMID 28123811
- [Background] Kerai S, Saxena KN, Taneja B. Post-caesarean analgesia: What is new? Indian J Anaesth. 2017 Mar;61(3):200-214. doi: 10.4103/ija.IJA_313_16. PMID 28405033
- [Background] Sultan P, Halpern SH, Pushpanathan E, Patel S, Carvalho B. The Effect of Intrathecal Morphine Dose on Outcomes After Elective Cesarean Delivery: A Meta-Analysis. Anesth Analg. 2016 Jul;123(1):154-64. doi: 10.1213/ANE.0000000000001255. PMID 27089000
- [Background] Al-Mustafa MM, Abu-Halaweh SA, Aloweidi AS, Murshidi MM, Ammari BA, Awwad ZM, Al-Edwan GM, Ramsay MA. Effect of dexmedetomidine added to spinal bupivacaine for urological procedures. Saudi Med J. 2009 Mar;30(3):365-70. PMID 19271064
- [Background] Qi X, Chen D, Li G, Huang X, Li Y, Wang X, Li Y. Comparison of Intrathecal Dexmedetomidine with Morphine as Adjuvants in Cesarean Sections. Biol Pharm Bull. 2016 Sep 1;39(9):1455-60. doi: 10.1248/bpb.b16-00145. Epub 2016 Jun 28. PMID 27349272
- [Background] Li XX, Li YM, Lv XL, Wang XH, Liu S. The efficacy and safety of intrathecal dexmedetomidine for parturients undergoing cesarean section: a double-blind randomized controlled trial. BMC Anesthesiol. 2020 Aug 3;20(1):190. doi: 10.1186/s12871-020-01109-4. PMID 32746864
- [Background] Bi YH, Wu JM, Zhang YZ, Zhang RQ. Effect of Different Doses of Intrathecal Dexmedetomidine as an Adjuvant Combined With Hyperbaric Ropivacaine in Patients Undergoing Cesarean Section. Front Pharmacol. 2020 Mar 20;11:342. doi: 10.3389/fphar.2020.00342. eCollection 2020. PMID 32265713
- [Background] Kim DJ, Ki YJ, Jang BH, Kim S, Kim SH, Jung KT. Clinically relevant concentrations of dexmedetomidine may reduce oxytocin-induced myometrium contractions in pregnant rats. Anesth Pain Med (Seoul). 2020 Oct 30;15(4):451-458. doi: 10.17085/apm.20036. PMID 33329848
- [Background] Cheng Q, Bi X, Zhang W, Lu Y, Tian H. Dexmedetomidine versus sufentanil with high- or low-concentration ropivacaine for labor epidural analgesia: A randomized trial. J Obstet Gynaecol Res. 2019 Nov;45(11):2193-2201. doi: 10.1111/jog.14104. Epub 2019 Sep 9. PMID 31502323
- [Background] Su F, Gastonguay MR, Nicolson SC, DiLiberto M, Ocampo-Pelland A, Zuppa AF. Dexmedetomidine Pharmacology in Neonates and Infants After Open Heart Surgery. Anesth Analg. 2016 May;122(5):1556-66. doi: 10.1213/ANE.0000000000000869. PMID 26218862
- [Background] Konakci S, Adanir T, Yilmaz G, Rezanko T. The efficacy and neurotoxicity of dexmedetomidine administered via the epidural route. Eur J Anaesthesiol. 2008 May;25(5):403-9. doi: 10.1017/S0265021507003079. Epub 2007 Dec 19. PMID 18088445
- [Background] Solanki SL, Goyal VK. Neuraxial dexmedetomidine: wonder drug or simply harmful. Anesth Pain Med. 2015 Mar 30;5(2):e22651. doi: 10.5812/aapm.22651. eCollection 2015 Apr. No abstract available. PMID 25866711
- [Background] Sanders RD, Sun P, Patel S, Li M, Maze M, Ma D. Dexmedetomidine provides cortical neuroprotection: impact on anaesthetic-induced neuroapoptosis in the rat developing brain. Acta Anaesthesiol Scand. 2010 Jul;54(6):710-6. doi: 10.1111/j.1399-6576.2009.02177.x. Epub 2009 Dec 9. PMID 20003127
- [Background] Celik F, Gocmez C, Kamasak K, Tufek A, Guzel A, Tokgoz O, Firat U, Evliyaoglu O. The comparison of neuroprotective effects of intrathecal dexmedetomidine and metilprednisolone in spinal cord injury. Int J Surg. 2013;11(5):414-8. doi: 10.1016/j.ijsu.2013.03.008. Epub 2013 Mar 28. PMID 23542594
- [Background] Crespo S, Dangelser G, Haller G. Intrathecal clonidine as an adjuvant for neuraxial anaesthesia during caesarean delivery: a systematic review and meta-analysis of randomised trials. Int J Obstet Anesth. 2017 Nov;32:64-76. doi: 10.1016/j.ijoa.2017.06.009. Epub 2017 Jun 27. PMID 28823524
- [Background] Engelman E, Marsala C. Efficacy of adding clonidine to intrathecal morphine in acute postoperative pain: meta-analysis. Br J Anaesth. 2013 Jan;110(1):21-7. doi: 10.1093/bja/aes344. Epub 2012 Sep 21. PMID 23002167
- [Background] Hassenbusch SJ, Gunes S, Wachsman S, Willis KD. Intrathecal clonidine in the treatment of intractable pain: a phase I/II study. Pain Med. 2002 Jun;3(2):85-91. doi: 10.1046/j.1526-4637.2002.02014.x. PMID 15102154
- [Background] Deer TR, Pope JE, Hayek SM, Lamer TJ, Veizi IE, Erdek M, Wallace MS, Grider JS, Levy RM, Prager J, Rosen SM, Saulino M, Yaksh TL, De Andres JA, Abejon Gonzalez D, Vesper J, Schu S, Simpson B, Mekhail N. The Polyanalgesic Consensus Conference (PACC): Recommendations for Intrathecal Drug Delivery: Guidance for Improving Safety and Mitigating Risks. Neuromodulation. 2017 Feb;20(2):155-176. doi: 10.1111/ner.12579. Epub 2017 Jan 2. PMID 28042914
- [Background] Schechtmann G, Lind G, Winter J, Meyerson BA, Linderoth B. Intrathecal clonidine and baclofen enhance the pain-relieving effect of spinal cord stimulation: a comparative placebo-controlled, randomized trial. Neurosurgery. 2010 Jul;67(1):173-81. doi: 10.1227/01.NEU.0000370249.41634.4F. PMID 20559103
- [Background] Remy-Neris O, Denys P, Bussel B. Intrathecal clonidine for controlling spastic hypertonia. Phys Med Rehabil Clin N Am. 2001 Nov;12(4):939-51, ix. PMID 11723871
- [Background] Teasell RW, Mehta S, Aubut JA, Foulon B, Wolfe DL, Hsieh JT, Townson AF, Short C; Spinal Cord Injury Rehabilitation Evidence Research Team. A systematic review of pharmacologic treatments of pain after spinal cord injury. Arch Phys Med Rehabil. 2010 May;91(5):816-31. doi: 10.1016/j.apmr.2010.01.022. PMID 20434623
- [Background] Chang E, Ghosh N, Yanni D, Lee S, Alexandru D, Mozaffar T. A Review of Spasticity Treatments: Pharmacological and Interventional Approaches. Crit Rev Phys Rehabil Med. 2013;25(1-2):11-22. doi: 10.1615/CritRevPhysRehabilMed.2013007945. PMID 25750484
- [Background] Pichot C, Longrois D, Ghignone M, Quintin L. [Dexmedetomidine and clonidine: a review of their pharmacodynamy to define their role for sedation in intensive care patients]. Ann Fr Anesth Reanim. 2012 Nov;31(11):876-96. doi: 10.1016/j.annfar.2012.07.018. Epub 2012 Oct 22. French. PMID 23089375
- [Background] Nedashkovsky EV, Sedykh SV, Zakurdaev EI. [USING A VISUAL ANALOGUE SCALE FOR ASSESSING THE SEVERITY OF PAIN SYNDROME AFTER CESAREAN SECTION, DEPENDING ON THE METHOD OF ANESTHESIA.]. Anesteziol Reanimatol. 2016 Sep;61(5):372-376. Russian. PMID 29489106
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Mizuno M, Fukunaga A, Washio K, Imamura S, Oda Y, Nishigori C. A visual analogue scale for itch and pain in 23 cases of cholinergic urticaria. J Eur Acad Dermatol Venereol. 2020 Sep;34(9):e493-e495. doi: 10.1111/jdv.16410. Epub 2020 May 28. No abstract available. PMID 32242985
- [Background] Craig D, Carli F. Bromage motor blockade score - a score that has lasted more than a lifetime. Can J Anaesth. 2018 Jul;65(7):837-838. doi: 10.1007/s12630-018-1101-7. Epub 2018 Mar 5. No abstract available. PMID 29508151
- [Background] Demumieux F, Ludes PO, Diemunsch P, Bennett-Guerrero E, Lujic M, Lefebvre F, Noll E. Validation of the translated Quality of Recovery-15 questionnaire in a French-speaking population. Br J Anaesth. 2020 Jun;124(6):761-767. doi: 10.1016/j.bja.2020.03.011. Epub 2020 Apr 15. PMID 32303379
- [Background] Bornstein E, Husk G, Lenchner E, Grunebaum A, Gadomski T, Zottola C, Werner S, Hirsch JS, Chervenak FA. Implementation of a Standardized Post-Cesarean Delivery Order Set with Multimodal Combination Analgesia Reduces Inpatient Opioid Usage. J Clin Med. 2020 Dec 22;10(1):7. doi: 10.3390/jcm10010007. PMID 33375192